CLINICAL TRIAL: NCT05691387
Title: Impact of the Active Cycle of Breathing Technique and Pursed Lip Breathing With TheraPep on People With Acute Episode of Chronic Obstructive Pulmonary Disease
Brief Title: Comparison of Active Cycle of Breathing Technique and Pursed Lip Breathing With TheraPep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Dr. Mohammad Abu Shaphe, Associate Professor, University of Jazan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: REC-44/06/445
Record Dates: First submitted 2023-01-10; First posted 2023-01-20 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Chronic Obstructive Pulmonary Disease Exacerbation
Keywords: chronic obstructive pulmonary disease; pursed lip breathing; active cycle breathing technique; airway clearance technique
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — phospholamban

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thera PEP (Experimental): Sitting comfortably, patients receiving Thera PEP will be told to place dental cotton swabs between their cheek and gum, and then under their tongue, to absorb saliva and prevent contamination of the collected sputum by the patient's own saliva. The diameter of the opening will be modified to achieve a ventilation rate of 1:4. The patient will be taught to take in a larger than normal breath but not fill the lungs to capacity in order to maintain a tight seal during exhalation. After completing ten PEP breaths, the patient will have the mouthpiece removed and be instructed to do two or three "puff" coughs. When secretions need to be brought up, a good cough will do the trick. During the duration of the treatment, which will last around thirty minutes, the patient will be asked to complete three cycles of ten breaths each.
  Interventions: Behavioral: Thera PEP
- ACBT and PLB (Active Comparator): On the day of the ACBT, the patient will be taught to place dental cotton swabs between the cheek and gum, as well as beneath the tongue, to absorb saliva and prevent contamination of the collected sputum by saliva. Throughout the treatment, the patient will be urged to maintain a comfortable sitting position. The patient will then be instructed to perform PLB at a normal tidal volume (for approximately 6 breaths), followed by 3-4 deep inspirations with relaxed exhalation (thoracic expansion exercise), and finally, another period of breathing control, i.e. PLB, followed by FET, i.e. a deep breath in and a huff cough, followed by a medium breath in and a huff cough again. Approximately thirty minutes will pass over the course of this session.
  Interventions: Behavioral: ACBT and PLB

INTERVENTIONS:
Behavioral: Thera PEP — Sitting comfortably, patients receiving Thera PEP will be told to place dental cotton swabs between their cheek and gum, and then under their tongue, to absorb saliva and prevent contamination of the collected sputum by the patient's own saliva. The diameter of the opening will be modified to achieve a ventilation rate of 1:4. The patient will be taught to take in a larger than normal breath but not fill the lungs to capacity in order to maintain a tight seal during exhalation. After completing ten PEP breaths, the patient will have the mouthpiece removed and be instructed to do two or three "puff" coughs. When secretions need to be brought up, a good cough will do the trick. During the duration of the treatment, which will last around thirty minutes, the patient will be asked to complete three cycles of ten breaths each.
  Other Names: ACBT and PLB
  Arms: Thera PEP
Behavioral: ACBT and PLB — On the day of the ACBT, the patient will be taught to place dental cotton swabs between the cheek and gum, as well as beneath the tongue, to absorb saliva and prevent contamination of the collected sputum by saliva. Throughout the treatment, the patient will be urged to maintain a comfortable sitting position. The patient will then be instructed to perform PLB at a normal tidal volume (for approximately 6 breaths), followed by 3-4 deep inspirations with relaxed exhalation (thoracic expansion exercise), and finally, another period of breathing control, i.e. PLB, followed by FET, i.e. a deep breath in and a huff cough, followed by a medium breath in and a huff cough again. Approximately thirty minutes will pass over the course of this session.
  Arms: ACBT and PLB

SUMMARY:
The purpose of this study is to investigate the short-term effects of two different breathing techniques (the active cycle breathing technique (ACBT) and the pursed lip breathing technique (PLB)) with Thera PEP® on the clearance of secretions and the oxygen saturation of individuals who have recently experienced an acute exacerbation of chronic obstructive pulmonary disease (COPD) in individuals who have recently experienced an acute exacerbation of COPD (COPD). Thirty patients will each have an acute COPD exacerbation seen on them, and then they will be randomly allocated to one of two groups (1. ACBT and PLB; 2. Thera PEP). Participants in a study employing a design known as a within-subject randomized crossover will be given the instruction to carry out each procedure on consecutive days as part of the study. In this study, the dependent variables will include blood pressure, heart rate, oxygen saturation (SpO2), respiratory rate, peak expiratory flow rate (PEFR), visual analog scale (VAS), sputum volume, and the breathlessness, cough, and sputum scale. In addition, the independent variables will include sputum volume (BCSC). The patient's desired course of treatment will also be taken into account. These dependent variables will be examined at three distinct moments in time: at the beginning of the study (the baseline), immediately after treatment, and thirty minutes after treatment has been completed.

DETAILED DESCRIPTION:
Methods:

There will be a total of thirty COPD patients recruited. Because of the rapid progression of their chronic obstructive pulmonary disease, these patients are going to need to be hospitalized. An acute exacerbation of COPD is suspected when there is an upper respiratory tract infection, a high temperature for no apparent reason, an increase in wheezing and coughing, or a rise in respiratory rate or heart rate above baseline. All of these symptoms are considered to be indications of an acute exacerbation of COPD. Co-morbidities, including but not limited to angina, indication for ventillatory support, neurological deficits, severe hemodynamic instability (including but not limited to cor pulmonale, cardiac arrhythmias, pulmonary embolism, pneumothorax, congestive heart failure, and GOLD stage IV: very severe COPD), and indication for ventilatory support will be used as exclusion criteria.

Interventions:

Individuals who will satisfy the inclusion and exclusion criteria will be given information regarding the two treatments (ACBT+PLB and PEP therapy to be offered by Thera PEP), and then they will be randomly randomized to either group (A or B) (A or B). Group A patients will get ACBT+PLB on day one of treatment, followed by PEP therapy using Thera PEP on day two. Treatment for patients in Group B will begin with PEP on Day 1, followed by ACBT+PLB on Day 2.

Sitting comfortably, patients receiving Thera PEP will be told to place dental cotton swabs between their cheek and gum, and then under their tongue, to absorb saliva and prevent contamination of the collected sputum by the patient's own saliva. The diameter of the opening will be modified to achieve a ventilation rate of 1:4. The patient will be taught to take in a larger than normal breath but not fill the lungs to capacity in order to maintain a tight seal during exhalation. After completing 10 PEP breaths, the patient will have the mouthpiece removed and be instructed to produce 2-3 "huff" coughs. When secretions need to be brought up, a good cough will do the trick. The patient will be instructed to do three sets of ten breaths each during the length of the therapy, which will last roughly thirty minutes in total. On the day of the ACBT, the patient will be instructed to place dental cotton swabs between the cheek and gum, as well as beneath the tongue, in order to absorb saliva and avoid the collected sputum from being tainted by the patient's own saliva. We'll want the patient to settle in for the duration of the procedure. After that, the patient will be given instructions to perform PLB at a normal tidal volume (for about 6 breaths), followed by 3-4 deep inspirations with relaxed exhalation (thoracic expansion exercise), and finally, another period of breathing control, i.e., PLB, followed by FET, i.e., a deep breath in and to do huff cough, followed by a medium breath in and again a huff cough. About thirty minutes will be spent in this procedure.

Outcome:

On day 0 (when no intervention is given), day 1 (at bedtime), and day 2, patients will be asked to fill out the sputum breathlessness cough scale (one of the dependent variables) (at bedtime). Besides the basics like pulse, blood pressure, and respiration rate, we'll also have a look at things like arterial oxygen saturation (SpO2), peak expiratory flow rate (PEFR), visual analog scale (VAS), and sputum volume to get a full picture of the patient's health (SV). Patients in both groups will be polled on which therapy modality they like best on Day 3.

Statistical analyses:

Data will be analyzed using SPSS for Windows, version 26. Treatment effects on the dependent variables will be analyzed using repeated-measures analysis of variance (ANOVA), with time as the within-subject component and the three measurements (baseline, posttest, and 30 minutes posttest) as the independent variables. Repeated-measures analysis will be used to examine correlations between participants, and a crossover layout will be used for variables that show statistical significance. The statistical study of the interaction between the period effect, the treatment period effect, and the treatment effect will be conducted using the independent-sample T-test. For the purposes of this research, a p value of 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients because of a rapid worsening of chronic obstructive pulmonary disease
* An upper respiratory tract infection
* a high temperature for no apparent reason
* an increase in wheezing and coughing, or
* a rise in respiratory rate or heart rate above baseline

Exclusion Criteria:

* Co-morbidities including but not limited to angina, indication for ventillatory support,
* neurological deficits,
* severe hemodynamic instability including but not limited to cor pulmonale, cardiac arrhythmias, pulmonary embolism, pneumothorax, congestive heart failure, and GOLD stage IV: very severe COPD; and
* indication for ventillatory support

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
blood pressure | Day 3
  A digital blood pressure monitor will be used. A tight-fitting arm cuff will be wrapped around the participant's upper arm before being inflated with air. Blood pressure that falls within the range of 90/60 mm Hg to 120/80 mm Hg is considered normal. Measurements of blood pressure will be taken before and after the intervention.
heart rate | Day 3
  Heart rate will be measured with a digital monitor while the person is supine at the beginning of the study and at the end of the intervention.
oxygen saturation (SpO2) | Day 3
  The oxygen saturation (SpO2) of the blood is a ratio of the amount of oxygen-carrying hemoglobin to the amount of total hemoglobin. Blood saturation levels of oxygen (SpO2) will be determined with the help of a pulse oximeter. The participant's finger will be positioned to receive the pulse oximeter. On the screen, you'll see a %. The usual range for this percentage, which measures how much oxygen hemoglobin can transport, is between 94% and 100%. This will be taken at baseline and end of intervention.
respiratory rate | Day 3
  The number of times in a minute that a person breathes is called their respiratory rate. An adult taking it easy should be breathing at a pace of 12-20 breaths per minute. It's abnormal to have a resting respiratory rate of less than 12 or more than 25 breaths per minute. This will be taken at baseline and end of intervention.
peak expiratory flow rate (PEFR) | Day 3
  A peak flow meter is a portable, hand-held instrument used to measure a person's maximal rate of exhalation (also known as peak expiratory flow or PEF). The test determines how much of an obstruction there is in the airways by measuring the airflow through the bronchi. Most of the time, people will use liters per minute (L/min) to describe their peak expiratory flow. When recording a patient's Peak Expiratory Flow Rate, the highest value from a set of three measurements will be used. This will be taken at baseline and end of intervention.
visual analog scale (VAS) | Day 3
  A visual analogue scale (VAS) is a line, typically 10 cm long, with word anchors at either end (such as "no pain" on the far left and "the most extreme pain imaginable" on the far right) to indicate a range of perceived discomfort. In order to indicate the level of pain experienced, the patient makes a mark on the line at the location that best represents their perception of that level of discomfort. A higher score indicate worst intensity of pain. This will be taken at baseline and end of intervention.
sputum volume | Day 3
  When the muco-ciliary escalator is working properly, the normal lung produces about 20 to 30 milliliters of mucus daily. When an excessive amount of mucus is formed in the airways and must be expectorated, this excess mucus is referred to as sputum. This will be taken at baseline and end of intervention.
the breathlessness, cough, and sputum scale (BCSC) | Day 3
  Patients will be requested to complete the sputum breathlessness cough scale (one of the dependent variables) on day 0 (when no intervention was given), at the end of day 1 (at bedtime), and at the end of day 2 (at bedtime).

CONTACTS AND LOCATIONS:
Overall Officials: Abu Shaphe, Principal Investigator — University of Jazan
Locations (1):
- Jazan University, Jizan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No